CLINICAL TRIAL: NCT00983814
Title: A Two-Period Trial (Open-Label and Randomized Placebo-Controlled Substitution) of Droxidopa Treatment in Adults With ADHD With Co-administration of Carbidopa
Brief Title: Study of Droxidopa Treatment in Adults With Attention Deficit Hyperactivity Disorder With Co-administration of Carbidopa
Acronym: ADD201
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chelsea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Droxidopa ADD201
Record Dates: First submitted 2009-09-23; First posted 2009-09-24 (Estimated); Results first posted 2024-04-18 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-03

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention Deficit Hyperactivity Disorder; ADHD; Adult ADHD; Adult Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Droxidopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Droxidopa+Carbidopa Open-Label (Experimental): 3 weeks of open label droxidopa (200, 400, or 600 milligrams [mg] three times daily [TID]) monotherapy followed by 3 weeks of droxidopa in combination with carbidopa (25 mg or 50 mg TID).
  Interventions: Drug: Droxidopa+Carbidopa
- Placebo Randomized Period (Placebo Comparator): 2 week double-blind period in which participants either continued to receive droxidopa+carbidopa treatment or placebo
  Interventions: Drug: Droxidopa+Carbidopa

INTERVENTIONS:
Drug: Droxidopa+Carbidopa — 3 weeks of open label droxidopa (L-dihydroxyphenylserine (L-DOPS)) (200, 400, or 600mgs TID) monotherapy followed by 3 weeks of droxidopa in combination with carbidopa (25mg or 50mg TID) followed by 2 weeks of double blind continued droxidopa+carbidopa or placebo
  Other Names: Droxidopa; L-threo-dihydroxyphenylserine; L-DOPS

SUMMARY:
Attention Deficit Hyperactivity Disorder (ADHD) is a neurobiological disorder characterized by lifelong issues of inattention, distraction, organizational difficulties, forgetfulness, restlessness, talking out of turn, difficulty waiting and interrupting others. ADHD is the second most common neuropsychiatric disorder affecting 4.4% of the United States (US) adult population, or between 8-9 million individuals.

Droxidopa (L-dihydroxyphenylserine (L-DOPS)) is a synthetic catecholamine which is converted to norepinephrine (NE) via decarboxylation, resulting in increased levels of NE centrally in the central nervous system (CNS) and peripherally. Co-treatment with carboxylase inhibitors, such as carbidopa, given with droxidopa, can increase the CNS levels of NE with greater crossing of the blood-brain barrier. Droxidopa has received orphan drug approval by the Food and Drug Administration (FDA) for the treatment of symptomatic neurogenic orthostatic hypotension in individuals with primary autonomic failure. The half-life of droxidopa is approximately 2-3 hours, resulting in administration three times daily.

DETAILED DESCRIPTION:
This will be a 12-week study of twenty enrolled participants with the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV) criteria adult ADHD (age 18-55), with a goal of completing twenty participants in the trial. The primary objective of this study is to determine the effect of droxidopa therapy on adult ADHD symptoms over the course of a six-week open-label titration period followed by a two-week double-blind, placebo-controlled period. The primary outcome measure will be changes from baseline in total score on the Adult ADHD Investigator Symptom Rating Scale (AISRS). Secondary measures will be changes in self-reported ADHD symptoms on the Adult ADHD Self-Report Scale (ASRS v1.1) and global impairment on the Clinician Global Impression Scale (CGI).

ELIGIBILITY:
Inclusion Criteria:

1. At the time of consent, are between the ages of 18-55, inclusive.
2. Meet DSM-IV criteria for ADHD as assessed by the Adult ADHD Clinician Diagnostic Scale (ACDS) v1.2.
3. Concomitant Axis I diagnoses that are allowed include social anxiety disorder or dysthymia which does not require treatment. Psychiatric co-morbidities will be diagnosed with the Structured Clinical Interview for DSM-IV Axis Disorders (SCID).
4. Must have a satisfactory medical assessment with no clinically significant abnormalities as determined by medical history, physical exam, electrocardiogram (ECG), and clinical laboratory testing.
5. Must be able to swallow capsules.
6. In the opinion of the investigator, the participant must understand and be able, willing and likely to fully comply with the study procedures and restrictions.
7. Must have given signed and dated informed consent in accordance with Good Clinical Practice (GCP) Guidelines.

Exclusion Criteria:

1. Lifetime or present history of bipolar or psychotic disorders, that in the investigator's opinion, interfere with the diagnosis and/or with the conduct of the study.
2. Uncontrolled comorbid major depressive disorder, anxiety disorder or dysthymia.
3. Women of childbearing potential who are not using a medically accepted contraception.
4. Sexually active males whose partner is a woman of child-bearing potential must agree to use condoms for the duration of the study and for 4 weeks after the last dose.
5. Women who are pregnant, breast feeding, or plan to become pregnant during the course of this study.
6. Clinically significant electrocardiogram or laboratory abnormalities at screening that are deemed exclusionary in the opinion of the Principal Investigator.
7. Participants taking any psychotropic medication on a regular basis. Participants will need to be free of all psychotropic medications (one week for psychostimulants, four weeks for all other medications), except for as needed (PRN) benzodiazepines or hypnotics. Allowed psychiatric co-morbidities include social anxiety disorder or dysthymia which does not require treatment.
8. Participants with any concurrent chronic or acute illness or unstable medical condition that could, in the opinion of the study physician, confound the results of safety assessments, increase risk to the participant or lead to difficulty complying with the protocol. Participants who have a history of mental retardation or severe learning disability will be excluded.
9. Participants who in the investigator's opinion meet any of the exclusionary criteria specified on the FDA label of either Droxidopa or carbidopa.
10. Have uncontrolled hypertension, defined as systolic blood pressure >140 millimeters of mercury (mmHg) and/or diastolic blood pressure >110 mmHg or use of ≥2 antihypertensive medications.
11. Known or suspected hypersensitivity to the study medication or any of its ingredients.
12. Have in the investigator's opinion any significant cardiac arrhythmia.
13. Any significant systemic, hepatic, cardiac or renal illness.
14. Diabetes mellitus or insipidus.
15. Have a history of closed angle glaucoma.
16. Have a known or suspected current malignancy. Participants with a history of cancer must be symptom- and treatment-free for at least 5 years prior to randomization, with the exception of participants with non-melanoma, non-invasive skin cancers (such as basal cell carcinoma), who should not have had an intervention or recurrence within one year of starting the study.
17. Participants with known gastrointestinal illness or other gastrointestinal disorder that may, in the investigator's opinion, affect the absorption of study drug.
18. In the investigator's opinion, have clinically significant abnormalities on clinical examination or laboratory testing.
19. In the investigator's opinion, are unable to adequately co-operate because of individual or family situation.
20. Are not able or willing to comply with the study requirements for the duration of the study.
21. Have participated in another clinical trial with an investigational agent (including named participant or compassionate use protocol) within 1 month before the start of the study.
22. Previous enrollment in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2009-10; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenard A Adler, M.D., Principal Investigator — VA New York Harbor Healthcare System/New York University Langone Medical Center
Locations (1):
- VA New York Harbor Healthcare System/New York University Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kessler RC, Adler L, Barkley R, Biederman J, Conners CK, Demler O, Faraone SV, Greenhill LL, Howes MJ, Secnik K, Spencer T, Ustun TB, Walters EE, Zaslavsky AM. The prevalence and correlates of adult ADHD in the United States: results from the National Comorbidity Survey Replication. Am J Psychiatry. 2006 Apr;163(4):716-23. doi: 10.1176/ajp.2006.163.4.716. PMID 16585449
- [Derived] Adler LA, Gorny SW. Pilot Study of Droxidopa With Carbidopa in Adults With ADHD. J Atten Disord. 2019 Jan;23(2):189-198. doi: 10.1177/1087054715580393. Epub 2015 Apr 23. PMID 25907673

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included 6 weeks of open-label and 2 weeks of double-blind treatment. A total of 20 participants were enrolled in the study. After 6 weeks of open-label treatment, participants were then randomized to either continue taking droxidopa+carbidopa or to receive placebo, for 2 weeks under double-blind conditions.
Groups:
- Droxidopa+Carbidopa: Open-Label: Participants received droxidopa monotherapy (titrated from 200 milligrams [mg] three times daily [TID] up to 600 mg TID orally depending on clinical response and tolerability) for 3 weeks followed by 3 weeks of fixed dose treatment with droxidopa (at the previously determined tolerable level) in conjunction with carbidopa (titrated from 25 mg TID to 50 mg TID orally, with potential step-down to 25 mg TID, depending on tolerability).
- Droxidopa+Carbidopa: Double-Blind: Participants received fixed dose treatment with droxidopa in conjunction with carbidopa (both at doses determined during open-label treatment) for 2 weeks.
- Placebo: Double-Blind: Participants received placebo matched capsules for droxidopa and carbidopa TID orally for 2 weeks.
Period: Open-Label (6 Weeks)
Arm/Group | Droxidopa+Carbidopa: Open-Label | Droxidopa+Carbidopa: Double-Blind | Placebo: Double-Blind
Started | 20 | 0 | 0
Received at Least 1 Dose of Study Drug | 2 | 0 | 0
Completed | 13 (2 participants withdrew after completing the open-label treatment and before entering the double-blind treatment.) | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0
Period: Double-Blind (2 Weeks)
Arm/Group | Droxidopa+Carbidopa: Open-Label | Droxidopa+Carbidopa: Double-Blind | Placebo: Double-Blind
Started | 0 | 6 | 5
Received at Least 1 Dose of Study Drug | 0 | 6 | 5
Completed | 0 | 6 | 4
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants, who went through screening and met all inclusion/exclusion criteria.
Groups:
- Droxidopa+Carbidopa: Open-Label Only: Participants received droxidopa monotherapy (titrated from 200 mg TID up to 600 mg TID orally depending on clinical response and tolerability) for 3 weeks followed by 3 weeks of fixed dose treatment with droxidopa (at the previously determined tolerable level) in conjunction with carbidopa (titrated from 25 mg TID to 50 mg TID orally, with potential step-down to 25 mg TID, depending on tolerability).
- Total: Total of all reporting groups
Arm/Group | Droxidopa+Carbidopa: Open-Label Only | Droxidopa+Carbidopa: Double-Blind | Placebo: Double-Blind | Total
Number analyzed (Participants) | 9 | 6 | 5 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 6 | 5 | 20
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: years] | 32 [23 to 53] | 37 [23 to 45] | 37 [21 to 40] | 34 [21 to 53]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 2 | 7
  Male | 5 | 5 | 3 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 0 | 1 | 0 | 1
  White | 6 | 2 | 5 | 13
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 5 | 20
Adult ADHD Investigator Symptom Report Scale (AISRS) Total Score [Mean (Standard Deviation); unit: units on a scale] — The AISRS is an 18-item validated investigator-administered instrument for the assessment of Attention Deficit Hyperactivity Disorder (ADHD) symptoms with an inattentive subscale (9 items) and a hyperactive-impulsive subscale (9 items). The severity of each of the items was rated on a 4-point scale (0-none, 1-mild, 2-moderate, 3-severe). The total score was the sum of the inattentive and hyperactive-impulsive subscales and ranged from 0 (none) to 54 (most severe). A higher score corresponded to a worse severity of ADHD.
  units on a scale | 35 (8.3) | 35 (7.9) | 32 (6.2) | 34 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Total AISRS Score at the End of Double-blind Treatment (Week 8)
Description: The AISRS is an 18-item validated investigator-administered instrument for the assessment of ADHD symptoms with an inattentive subscale (9 items) and a hyperactive-impulsive subscale (9 items). The severity of each of the items was rated on a 4-point scale (0-none, 1-mild, 2-moderate, 3-severe). The total score was the sum of the inattentive and hyperactive-impulsive subscales and ranged from 0 (none) to 54 (most severe). A higher score corresponded to a worse severity of ADHD.
Time Frame: Baseline, Week 8
Population: ITT population included all enrolled participants, who went through screening and met all inclusion/exclusion criteria. Missing data were imputed using the last observation carried forward (LOCF) method. Only participants who received the double-blind treatment were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa+Carbidopa: Double-Blind | Placebo: Double-Blind
Number analyzed (Participants) | 6 | 5
units on a scale | -17 (10.4) | -17 (4.1)

2. Secondary Outcome: Change From Baseline in Adult ADHD Self-Report Scale (ASRS) v1.1 Total Score at the End of Double-blind Treatment (Week 8)
Description: ASRS is a validated self-administered, instrument for the assessment of ADHD symptoms. It comprised of 18 items, which were rated by the participant on a 5-point scale (0=never, 1=rarely, 2=sometimes, 3=often, 4=very often). Total ASRS score was the sum of the ordinal response values for the 18 ASRS questions and ranged from 0 (never) to 72 (very often). A higher score corresponded to a worse severity of ADHD.
Time Frame: Baseline, Week 8
Population: ITT population included all enrolled participants, who went through screening and met all inclusion/exclusion criteria. Missing data were imputed using the LOCF method. Only participants who received the double-blind treatment were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa+Carbidopa: Double-Blind | Placebo: Double-Blind
Number analyzed (Participants) | 6 | 5
units on a scale | -15 (5.1) | -19 (8.6)

3. Secondary Outcome: Change From Baseline in Global Impairment on the Clinician Global Impression (CGI) Scale at the End of Double-blind Treatment (Week 8)
Description: 7-point clinician-rated scale assessing global severity of ADHD ranging from Normal (1), Borderline (2), Mild (3), Moderate (4), Marked (5), Severe (6), to Extremely Severe (7) in functional impairment.
Time Frame: Baseline, Week 8
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Droxidopa+Carbidopa: Double-Blind | Placebo: Double-Blind
Number analyzed (Participants) | 6 | 5
units on a scale | -1 (1.2) | -1 (0.9)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 12
Description: Safety population included all enrolled participants who received at least one dose of study drug.
Groups:
- Droxidopa+Carbidopa: Open-Label: Participants received droxidopa monotherapy (titrated from 200 mg TID up to 600 mg TID orally depending on clinical response and tolerability) for 3 weeks followed by 3 weeks of fixed dose treatment with droxidopa (at the previously determined tolerable level) in conjunction with carbidopa (titrated from 25 mg TID to 50 mg TID orally, with potential step-down to 25 mg TID, depending on tolerability).
Arm/Group | Droxidopa+Carbidopa: Open-Label | Droxidopa+Carbidopa: Double-Blind | Placebo: Double-Blind
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 14/20 | 1/6 | 0/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Droxidopa+Carbidopa: Open-Label (N=20) | Droxidopa+Carbidopa: Double-Blind (N=6) | Placebo: Double-Blind (N=5)
Headache (Nervous system disorders) | 5 (5) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 5 (5) | 0 (0) | 0 (0)
Depressed Mood (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Insomnia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No